CLINICAL TRIAL: NCT01312844
Title: A Pilot Study of the Use of IV Scopolamine to Augment the Efficacy of Electroconvulsive Therapy (ECT)
Brief Title: A Study of the Use of IV Scopolamine to Augment the Efficacy of Electroconvulsive Therapy (ECT)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This was an inpatient study, but PI left inpatient service at MGH
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, John D. Matthews, Principal Investigator, Assistant Professor of Psychiatry, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009P002288
Record Dates: First submitted 2010-05-04; First posted 2011-03-11 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Scopolamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Scopolamine (Experimental): Patients receiving IV scopolamine at ECT treatment
  Interventions: Drug: Scopolamine
- Placebo (Placebo Comparator): Patients receiving IV placebo at ECT treatment
  Interventions: Drug: Scopolamine

INTERVENTIONS:
Drug: Scopolamine — Those receiving active drug will receive scopolamine 4mcg/kg IV with each treatment, until completion of ECT

SUMMARY:
The primary purpose of this study is to assess the ability of scopolamine to improve the antidepressant effects of ECT and to determine whether scopolamine will shorten the time to response and remission for patients receiving ECT.

The hypothesis are:

1. Patients receiving ECT plus scopolamine will have greater improvement in depression symptoms than those receiving ECT plus placebo.
2. Patients receiving scopolamine in addition to ECT will require fewer ECT treatments to obtain response/remission compared to the group receiving ECT plus placebo.
3. Time to response and to remission in the scopolamine group will be significantly shorter compared to ECT alone.

DETAILED DESCRIPTION:
Electroconvulsive therapy (ECT) is a highly effective treatment for severe major depression. It has been estimated that approximately 10 percent of all patients admitted to the hospital for treatment of major depressive disorder receive ECT.

However, not all patients who receive ECT respond, and of those who do, not all achieve remission. Furthermore, while there is a wide range in the number of ECT treatments done among all people with depression, the average is approximately eight treatments. Because treatments are usually done three times per week (Monday, Wednesday, and Friday), the minimal length of stay for the average person receiving inpatient ECT is typically greater than two weeks.

Finally, ECT is not without risk, and every round of ECT incurs additional risk of not just the treatment itself, but also the risks of general anesthesia. Thus, although ECT is a robust mode of treatment for Major Depressive Disorder (MDD), there remains a need for improved treatment efficacy and speed of onset. Improving the efficacy of ECT would not only benefit individuals with MDD, but also have far-reaching effects for the health care system as it could impact the cost and resources utilized.

Ideally, an agent could be added to augment the effect of ECT, both in terms of efficacy as well as speed of onset. In 2006, Furrey et al, reported the rapid antidepressant effect of the antimuscarinic drug, scopolamine, delivered parenterally. Significant antidepressant effect was found after the first scopolamine administration. The improvement was reported immediately following the first IV administration, increased across all treatments, and was sustained into the placebo crossover period.

Scopolamine is an anticholinergic muscarinic agent, with activity in the CNS and pilot data to suggest a significant impact on rapidly improving depressive symptoms in patient with MDD, when administered IV. Thus, it serves as a reasonable choice to augment the effects of ECT in the treatment of patients with MDD.

Primary Aim 1) Assess the ability of scopolamine to augment the antidepressant effects of ECT.

Hypothesis 1a: Patients receiving ECT plus scopolamine will have significantly greater mean improvement on total HAM-D score between baseline and endpoint than those receiving ECT plus placebo.

Hypothesis 1b: Patients receiving scopolamine in addition to ECT will require fewer mean ECT treatments to obtain response/remission compared to the group receiving ECT plus placebo.

Primary Aim 2) Evaluate the hypothesis that scopolamine will shorten the time to response and remission for patients receiving ECT.

Hypothesis 2: Time to response and to remission in the Scopolamine group will be significantly shorter compared to ECT alone.

Secondary Aim: Provide evidence for the tolerability of intravenous scopolamine administered during ECT.

Hypothesis 3a: There will be no between group difference (between ECT plus scopolamine vs ECT plus placebo) in mean number of ECT sessions withheld due to cognitive impairment (as determined by attending psychiatrist).

Hypothesis 3b: There will be no between group differences (between ECT plus scopolamine vs ECT plus placebo) with regards to the mean number of moderate to severe side effects.

Hypothesis 3c: There will be no significant difference between the scopolamine plus ECT group and the placebo plus ECT group on mean levels of physiological measures of ECT including: heart rate, blood pressure, seizure length, duration of muscle paralysis, duration of asystole, and energy need to induce seizure.

Exploratory Analyses: we will assess whether the scopolamine plus ECT group will have a shorter average length of stay on the inpatient psychiatric unit compared to those receiving ECT plus placebo.

We will also assess whether the scopolamine plus ECT group will have significant differences in the cognitive measures at endpoint compared to those receiving ECT plus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 18-50 (inclusive)
* DSM-IV diagnosis of Major Depressive Disorder (MDD), without psychotic features, and a HAM-D-17 score of 18 or higher
* Female subjects must be postmenopausal, surgically sterile, or, if of child-bearing age, using double-barrier contraceptive method or prescription oral contraceptives (e.g. estrogen-progestin combinations), contraceptive implants (e.g. NorplantTM, DepoProveraTM, or transdermally delivered contraceptives (Ortho EvraTM) before entry and throughout the study; and have a negative urine b-HCG pregnancy test at screening.

Exclusion Criteria:

1. Substance use disorder active use within the last 6 months (per assessment using SCID)
2. Organic mental disorders
3. Seizure disorders
4. Unstable physical disorder or physical disorder judged to significantly affect the central nervous system function
5. Heart block
6. Pre-existing sick-sinus
7. Chronic treatment with beta blockers
8. Any cardiac arrhythmia
9. Hypotension
10. Coronary artery disease
11. Liver and renal function impairment
12. Urge incontinence or prostatic hypertrophy
13. Colitis
14. Crohn's disease
15. GI motility disorders
16. Asthma
17. COPD
18. Treatment with anti-cholinergic and cholinomimetic medications
19. Contraindications to scopolamine including hypersensitivity to scopolamine, other belladonna alkaloids, and/or any component of the formulation
20. Wide and narrow angle glaucoma
21. Acute hemorrhage
22. Paralytic ileus
23. Myasthenia gravis
24. Patients on belladonna, belladonna alkaloids, cisapride, or potassium chloride

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2010-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D Matthews, MD, Principal Investigator — Massachusetts General Hospital; David Abramson, MD, Principal Investigator — Massachusetts General Hospital; Maurizio Fava, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Scopolamine | Placebo
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Scopolamine | Placebo | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.25 (8.62) | 56.67 (21.78) | 51.86 (14.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Ham D 17 Scores
Description: Change in Ham D 17 scores measured by the difference between baseline HAM D score and HAM D score at last ECT administration. The HAM D 17 measures severity of depression with 52 being most severe and 0 being no depression. A negative change score refers to a decrease in HAM D score, while a positive change score would refer to an increase in HAM D score.
Time Frame: At the time of ECT completion (about 2 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scopolamine | Placebo
Number analyzed (Participants) | 4 | 3
units on a scale | -17.50 (10.47) | -14.00 (11.00)

2. Primary Outcome: Time to Response for Patients Receiving ECT
Description: The number of days between baseline HAM D score and HAM D score showing response (defined as a HAM D score less than half of baseline). If patients HAM D score rose above this marker at any point in the study, they were not considered as responding.The HAM D 17 measures severity of depression with 52 being most severe and 0 being no depression. .
Time Frame: Duration of ECT treatment (usually 2 weeks)
Population: Only 3 (out of 4) Scopolamine patients and 2 (out of 3) placebo patients reached response
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Scopolamine | Placebo
Number analyzed (Participants) | 3 | 2
days | 8.33 (3.21) | 5.00 (1.41)

3. Primary Outcome: Number of ECT Treatments Received to Achieve Response/Remission
Description: The number of ECT treatments needed to achieve response (defined as a HAM D score less than half of baseline) and remission (defined as a HAM D score of less than 8). If patients HAM D score rose above these markers at any point in the study, they were not considered as responding or remitting.The HAM D 17 measures severity of depression with 52 being most severe and 0 being no depression.
Time Frame: Duration of ECTtreatment (usually 2 weeks)
Population: Only 3 (out of 4) Scopolamine patients and 2 (out of 3) placebo patients reached response and remission.
Measure: Mean (Standard Deviation); unit: # of ECT administrations
Arm/Group | Scopolamine | Placebo
Number analyzed (Participants) | 3 | 2
# of ECT administrations
  # of ECT administrations to response | 2.33 (2.21) | 2.50 (0.71)
  # of ECT administrations to remission | 10.00 (3.46) | 6.50 (0.71)

4. Secondary Outcome: Number of ECT Treatments Withheld Due to Cognitive Impairment
Description: The number of ECT treatments withheld during the course of the study due to cognitive impairment. In these cases, the participant would still be enrolled in the study but have a reduced # of ECTs. This outcome measure does not include patients who withdrew from the study.
Time Frame: Duration of ECT treatment (usually 2 weeks)
Measure: Mean (Standard Deviation); unit: ECT Treatments withheld
Arm/Group | Scopolamine | Placebo
Number analyzed (Participants) | 3 | 3
ECT Treatments withheld | 0 (0) | 0 (0)

5. Secondary Outcome: The Mean Number of Moderate to Severe Side Effects
Description: The mean number of adverse events classified as moderate to severe.
Time Frame: Duration of ECT treatment (usually 2 weeks)
Measure: Mean (Standard Deviation); unit: number of side effects
Arm/Group | Scopolamine | Placebo
Number analyzed (Participants) | 4 | 3
number of side effects | .75 (1.5) | 0 (0)

6. Secondary Outcome: The Mean Levels of Physiological Measures of ECT (Blood Pressure)
Description: Blood pressure was taken immediately post ECT administration at each ECT visit. We averaged Blood pressure for each participant at each ECT administration. The reported mean refers to the average among all participants in each group.
Time Frame: Duration of ECT treatment (usually 2 weeks)
Population: Missing vitals forms for one participant in Scopolamine group (n=4), only reported data for 3 participants in Scopolamine group
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Scopolamine | Placebo
Number analyzed (Participants) | 3 | 3
mmHg
  Systolic blood pressure immediately post ECT | 170.35 (37.88) | 131.05 (27.57)
  Diastolic Blood Pressure Immediately Post ECT | 87.41 (16.92) | 78.80 (16.61)

7. Secondary Outcome: The Mean Levels of Physiological Measures of ECT (Heart Rate)
Description: Heart rate was taken immediately post ECT administration at each ECT visit. We averaged heart rate for each participant at each ECT administration. The reported mean refers to the average among all participants in each group.
Time Frame: Duration of ECT treatment (usually 2 weeks)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Scopolamine | Placebo
Number analyzed (Participants) | 3 | 3
Beats per minute | 69.24 (11.45) | 86.20 (15.62)

8. Secondary Outcome: The Mean Levels of Physiological Measures of ECT (Seizure Duration)
Description: Mean duration in seconds of the seizure induced by ECT for each participant at each ECT administration they received.The reported mean refers to the average among all participants in each group.
Time Frame: Duration of ECT treatment (usually 2 weeks)
Population: Missing ECT forms for one participant in Scopolamine group (n=4), only reported data for 3 participants in Scopolamine group
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Scopolamine | Placebo
Number analyzed (Participants) | 3 | 3
seconds | 30.25 (7.77) | 31.89 (10.56)

9. Secondary Outcome: The Mean Levels of Physiological Measures of ECT (Energy Needed)
Description: Mean energy needed to induce the seizure for each participant at each ECT administration they received. The reported mean refers to the average among all participants in each group.
Time Frame: Duration of ECT treatment (usually 2 weeks)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: joules
Arm/Group | Scopolamine | Placebo
Number analyzed (Participants) | 3 | 3
joules | 73.83 (31.12) | 67.06 (30.02)

ADVERSE EVENTS:
Arm/Group | Scopolamine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/3
Other Adverse Events (participants affected / at risk) | 1/4 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Scopolamine (N=4) | Placebo (N=3)
Recent memory loss (Nervous system disorders) | 1 (1) | 0 (0)
Agitation requiring restraint (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Scopolamine (N=4) | Placebo (N=3)
Deja vu / confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Hypoxia event (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes